CLINICAL TRIAL: NCT06060223
Title: The Effect of Teach Back Method on Symptom Control, Treatment Compliance and Self-Care Behaviors in Individuals With Heart Failure
Brief Title: Teach Back Method in Individuals With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-TG-777
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: patient; education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach Back Method (Experimental): Training and consultancy services based on the teach-back method will be provided to individuals in the training group using the "Heart Failure Training Guide" in the form of 3 follow-ups in the cardiology clinic and telephone counseling. Telephone interviews were conducted by the researcher in the first week after discharge, it will be held in the first month and 3rd month. In addition, patients will receive counseling by calling the researcher if necessary.
  Interventions: Other: Teach Back Method
- Control (No Intervention): Patients in the control group will participate in standard educational practices implemented in the clinic.Patients will be contacted by phone 3 months after discharge. Data collection forms will be applied as a final test.

INTERVENTIONS:
Other: Teach Back Method — Training and consultancy services based on the teach-back method will be provided to individuals in the training group using the "Heart Failure Training Guide" in the form of 3 follow-ups in the cardiology clinic and telephone counseling. Telephone interviews were conducted by the researcher in the first week after discharge, it will be held in the first month and 3rd month. In addition, patients will receive counseling by calling the researcher if necessary.
  Arms: Teach Back Method

SUMMARY:
This study will be conducted to determine the effect of the training given to indivuduals with heart failure by teach back method on their symptom control, adherence to treatment and self care behaviours.

DETAILED DESCRIPTION:
İntroduction: At least 40 million individuals worldwide live with heart failure. Although it is progressive, heart failure symptoms can be controlled through pharmacological treatment and self-care practices. The aim of heart failure treatment is to improve the quality of life of patients, prolong their lifespan, and prevent the progression of symptoms of the disease and re-admission to the hospital. Heart failure guidelines state that patient education and post-discharge follow-up are necessary for successful management of symptoms.

Purpose:This study will be conducted to determine the effect of the training given to indivuduals with heart failure by teach back method on their symptom control, adherence to treatment and self care behaviours.

Method:This study will be conducted using a randomized controlled research design. The research sample will consist of 58 with heart failure in the cardiology department of a training and research hospital. Research data will be collected using introductory information form, the Morsky Treatment Compliance Scale, European Heart Failure Self-Care Behavior Scale-12, Heart Failure Symptom Status Scale. Training and consultancy services based on the teach-back method will be provided to individuals in the training group using the "Heart Failure Training Guide" in the form of 3 follow-ups in the cardiology clinic and telephone counseling. Telephone interviews were conducted by the researcher in the first week after discharge, it will be held in the first month and 3rd month. In addition, patients will receive counseling by calling the researcher if necessary. After the patients are discharged, they will be called 1 week later, at the end of the 1st month and at the end of the 3rd month, and training will be repeated and counseling will be provided in line with the issues needed. Research posttest data will be collected 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with heart failure at least 6 months ago
* Individuals who speak and understand Turkish
* Able to communicate by phone
* İndividuals who can read and write
* Those who gave consent to participate in the research

Exclusion Criteria:

* under 18 years old
* Patients with cognitive dysfunction
* Those with neuro-psychiatric disease
* Those who did not consent to participate in the research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Morsky Treatment Compliance Scale (MTUÖ-8) | 3 months
  The scale consists of seven yes/no closed-ended questions with two options and one closed-ended question with five options. 1 point is given for answering no to questions one, two, three, four, six and seven, and 1 point is given for answering yes to question five. The eighth question consists of a multiple choice question called Likert type.A high score from the scale indicates high compliance with treatment.
European Heart Failure Self-Care Behavior Scale-12 | 3 months
  The scale applied to measure the self-care behaviors of patients with heart failure has been determined as a scale that provides results in a short time, does not require separate training, and can be applied by the patients themselves. Identifying symptoms related to heart failure such as edema, respiratory distress, and fatigue; It is a Likert-type scale consisting of 12 questions that measures self-care assessment actions such as regular use of medications for these symptoms, fluid and salt restriction, communication with healthcare personnel, and weight monitoring.A high total score indicates low self-care, a low score indicates high self-care.
Heart Failure Symptom Status Scale | 3 months
  Developed by et al. aimed to evaluate the presence, frequency and severity of seven main symptoms, such as dyspnea during the day, dyspnea while lying down, fatigue, angina, edema, sleep problems, dizziness or loss of balance, which are the most common in HF patients, and to what extent each of them affects the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Neşe Uysal, Study Director — Amasya U
Locations (1):
- Amasya University, Merkez, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No